CLINICAL TRIAL: NCT03297944
Title: Alprazolam and Simulated Driving Performance: Next Day Effects
Brief Title: Sedative-Anxiolytic Effects on Simulated Driving Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marion Coe (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Marion Coe, Doctoral Candidate, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-0260-F6A; R36DA043714-01A1 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Psychomotor Impairment
MeSH Terms: conditions — Psychomotor Disorders | interventions — Alprazolam; Zolpidem

STUDY DESIGN:
Masking Description: Participants and outcomes assessors were masked with respect to each individual intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Experimental): All participants received each intervention with alprazolam, zolpidem and placebo.
  Interventions: Drug: Alprazolam 2mg (2ALP/PLC); Drug: Alprazolam 1mg (1ALP/PLC); Drug: Alprazolam 0.5mg (0.5ALP/PLC); Drug: Zolpidem 10mg (ZOL/PLC); Drug: Placebo (PLC/PLC); Drug: Alprazolam 1mg (PLC/ALC)

INTERVENTIONS:
Drug: Alprazolam 2mg (2ALP/PLC) — 2mg alprazolam administered at night, placebo administered in the morning.
Drug: Alprazolam 1mg (1ALP/PLC) — 1mg alprazolam administered at night, placebo administered in the morning.
Drug: Alprazolam 0.5mg (0.5ALP/PLC) — 0.5mg alprazolam administered at night, placebo administered in the morning.
Drug: Zolpidem 10mg (ZOL/PLC) — 10mg alprazolam administered at night, placebo administered in the morning.
Drug: Placebo (PLC/PLC) — Placebo administered at night, placebo administered in the morning.
Drug: Alprazolam 1mg (PLC/ALC) — Placebo administered at night, 1mg alprazolam administered in the morning.

SUMMARY:
This study evaluates the effect of anxiety drugs taken at night on the ability to drive a car the next day. Participants will receive alprazolam, placebo, or zolpidem at night before bed or in the morning before using a driving simulator to assess impairment.

ELIGIBILITY:
Inclusion Criteria:

* valid driver's license
* english-speaking and literate

Exclusion Criteria:

* using daily medication for chronic condition
* acute narrow angle glaucoma
* previous adverse experience with study drugs
* experiences motion sickness in response to driving simulator
* BMI > 30
* women who are pregnant, lactating, or planning on becoming pregnant
* regular use of tobacco products
* current substance use disorder
* clinically significant ECG
* current ongoing psychiatric disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Coe, Principal Investigator — University of Kentucky
Locations (1):
- Center on Drug and Alcohol Research, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roszkowski SC, Babalonis S, Coe MA, Nuzzo PA, Lofwall MR, Fanucchi LC, Walsh SL. Residual next-day effects of alprazolam on psychomotor performance and simulated driving in healthy normal adults. Exp Clin Psychopharmacol. 2025 Apr;33(2):178-188. doi: 10.1037/pha0000746. Epub 2024 Nov 14. PMID 39541522

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 15 participants received every intervention.
Groups:
- All Participants: All participants received all six interventions; combinations of placebo (PLC), alprazolam (ALP) or zolpidem (ZOL).
Period: Overall Study
Arm/Group | All Participants
Started | 15
2ALP/PLC | 15
1ALP/PLC | 15
0.5ALP/PLC | 15
ZOL/PLC | 15
PLC/PLC | 15
PLC/ALP | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All 15 participants received each intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.53 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation of Lane Position (SLDP)
Description: Lane deviation (swerving) on a driving simulator. This is measured as the distance (cm) the driver deviates from the lane.
Time Frame: 16 hours
Population: All 15 participants received each intervention.
Measure: Mean (Full Range); unit: distance (cm)
Groups:
- All Participants: All participants received all 6 interventions.
Arm/Group | All Participants
Number analyzed (Participants) | 15
distance (cm)
  2ALP/PLC | 40.08 [28.1 to 68.1]
  1ALP/PLC | 37.28 [28.0 to 54.9]
  0.5ALP/PLC | 36.06 [27.6 to 53.7]
  ZOL/PLC | 37.61 [28.3 to 65.6]
  PLC/PLC | 36.30 [29.7 to 58.9]
  PLC/ALP | 40.72 [28.5 to 68.7]

ADVERSE EVENTS:
Time Frame: 16 hours
Groups:
- 2ALP/PLC: 2mg Alprazolam administered at night, placebo administered in the morning
  Alprazolam: 0.5 to 2mg administered at night or in the morning
- 1ALP/PLC: 1mg Alprazolam administered at night, placebo administered in the morning
  Alprazolam: 0.5 to 2mg administered at night or in the morning
- 0.5ALP/PLC: 0.5mg Alprazolam administered at night, placebo administered in the morning
  Alprazolam: 0.5 to 2mg administered at night or in the morning
- ZOL/PLC: 10mg Zolpidem administered at night, placebo administered in the morning
  Zolpidem: 10mg administered at night or in the morning
- PLC/PLC: Placebo administered at night, placebo administered in the morning
  Placebo: placebo administered at night and/or in the morning
- PLC/ALP: Placebo administered at night, 1mg alprazolam administered in the morning
  Alprazolam: 0.5 to 2mg administered at night or in the morning
Arm/Group | 2ALP/PLC | 1ALP/PLC | 0.5ALP/PLC | ZOL/PLC | PLC/PLC | PLC/ALP
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/15 | 2/15 | 0/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2ALP/PLC (N=15) | 1ALP/PLC (N=15) | 0.5ALP/PLC (N=15) | ZOL/PLC (N=15) | PLC/PLC (N=15) | PLC/ALP (N=15)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach Ache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03297944/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03297944/Prot_SAP_001.pdf